CLINICAL TRIAL: NCT04183569
Title: Identification Predictive Markers of Immunochemotherapy Response to the Primary Cutaneous Diffuse Large B Cell Lymphoma by Transcriptomic Proteomics and Mutational Analysis
Brief Title: Identification Predictive Markers of Immunochemotherapy Response to the Primary Cutaneous Diffuse Large B Cell Lymphoma
Acronym: PROTEOM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2018/78
Record Dates: First submitted 2019-11-28; First posted 2019-12-03 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Lymphoma, Large B-Cell, Diffuse
Keywords: Proteomic; Mutations; Predictive marker; Rituximab-polychemotherapy; Integrative bioinformatics tool
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Base Sequence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — skin biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary diffuse cutaneous B-cell lymphoma, leg type: Cohort of 32 patients LBC-TJ treated with R-chemotherapy for which data collection was carried out in homogeneous and prospectively followed according to international standards through RCP monthly cutaneous lymphomas managed by Professor Beylot-Barry and inclusion of cases in the national database of rare cancer network French Study Group of Cutaneous Lymphomas in Bordeaux managed by Prof. Beatrice Vergier.
  Interventions: Other: Sequencing RNA.

INTERVENTIONS:
Other: Sequencing RNA. — RNA-seq, central pivot between genomics and proteomics allows to make the connection between the observed mutations and alteration of protein expression with the identification and quantification of RNA. Thus, we can attest to the expression of mutations identified on DNA, protein and understand whether deregulation is linked to dysregulation of transcription or post-translational modification

SUMMARY:
The study is performed on a single-center retrospective cohort of 32 patients LBC-TJ treated with R-chemotherapy for which data collection was carried out in homogeneous and prospectively followed according to international standards through RCP monthly cutaneous lymphomas managed by Professor Beylot-Barry and inclusion of cases in the national database of rare cancer network French Study Group of Cutaneous Lymphomas in Bordeaux managed by Prof. Beatrice Vergier. Fourteen patients responded to the R-PCT against 18 non-responders, 14 patients for whom we have the sample to recidivism.

DETAILED DESCRIPTION:
The objective is to identify predictive biomarkers of response to R-chemotherapy and understand what genomic markers, transcriptomic or proteomic would identify those patients ahead. This would ultimately help to identify whether dysregulated biological pathway could be targeted specifically among patients with personalized treatment.

Like its counterpart systemic Lymphoma Diffuse large B cell, the sequential analysis of the same patient at diagnosis and relapse can also identify candidate genes and biological pathways involved in recurrence and help to design new therapeutic strategies.

Another objective is ultimately the development of an integrative bioinformatics tool for anticipating the therapeutic response. The tumor model used is certainly a rare cancer but prototypical ABC lymphomas allowing access to relapse hardware and relative homogeneity that will allow a study of a smaller number of cases for the development of correlations models genomics / proteomics. This is a pivotal project integrating proteomic data and Molecular Biology (mutation, expression) based on the pooling of skills of clinical teams, biological and bioinformatics to validate a predictive model for treatment response able to integrate prognostic markers known as TNM the dual expression MYC / BCL2 and forward to predict the therapeutic response using this modeling by CBIB. We would then validate the model established in this series of training on a range of national validation as part of an observational study with GFELC (Groupe Français d'Etude des Lymphomes Cutanés).

ELIGIBILITY:
* Patients LBC-TJ
* Treated with R-chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients LBC-TJ treated with R-chemotherapy for which data collection was carried out in homogeneous and prospectively followed according to international standards through RCP monthly cutaneous lymphomasmanaged by Professor Beylot-Barry and inclusion of cases in the national database of rare cancer network French Study Group of Cutaneous Lymphomas in Bordeaux managed by Prof. Beatrice Vergier.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Describe of mutations in genes | day1
  To characterize the tumours, a sequencing of dedicated lymphopanel targeting the most frequently altered genes in large B-cell lymphomas was performed. Several highly recurrent mutations of MYD88, PIM1, CD79B and MYC, as well as CDKN2A, BLIMP1 and TNFAIP3 deletions were detected per patient leading to the putative deregulation of several biological pathways. These sequencing data have evidenced the genetic diversity and complexity of PCLBCL, LT mutational landscape.

CONTACTS AND LOCATIONS:
Overall Officials: Audrey GROS, PharmD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Service de Biologie des Tumeurs et Tumorothèque, Pessac, France

IPD SHARING:
Plan to Share IPD: No